CLINICAL TRIAL: NCT01102673
Title: A Phase 1 Placebo-Controlled Trial to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Food Effect of Single Escalating Oral Doses of PF-04991532 in Healthy Adult Subjects
Brief Title: Single Dose Study of PF-04991532 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: B2611001
Record Dates: First submitted 2010-04-12; First posted 2010-04-13 (Estimated); Last update posted 2010-08-05 (Estimated); Status verified 2010-08

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders
Keywords: phase 1; safety and tolerability; PK; T2DM; type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders | interventions — 6-(3-cyclopentyl-2-(4-(trifluoromethyl)-1H-imidazol-1-yl)propanamido)nicotinic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04991532 (Experimental): This will be a crossover study with 2 cohorts and an interleaving design with placebo substitution. The study will be conducted over 4 treatment periods in Cohort 1 (n=9) and over 3 treatment periods in Cohort 2 (n=9). Six subjects will be allocated to receive PF-04991532 and three subjects will be allocated to receive placebo treatment during each dosing period, except for the 4th period of Cohort 1. The 4th period of Cohort 1 will be dedicated to assess the effect of food on PF-04991532 PK parameters at one of the doses previously tested in Cohort 1; hence all 9 subjects will be dosed with PF-04991532 in an open-label fashion. A washout period of at least 7 days will occur between each dose.
  Interventions: Drug: PF-04991532
- Placebo (Placebo Comparator): This will be a crossover study with 2 cohorts and an interleaving design with placebo substitution. The study will be conducted over 4 treatment periods in Cohort 1 (n=9) and over 3 treatment periods in Cohort 2 (n=9). Six subjects will be allocated to receive PF-04991532 and three subjects will be allocated to receive placebo treatment during each dosing period, except for the 4th period of Cohort 1. The 4th period of Cohort 1 will be dedicated to assess the effect of food on PF-04991532 PK parameters at one of the doses previously tested in Cohort 1; hence all 9 subjects will be dosed with PF-04991532 in an open-label fashion. A washout period of at least 7 days will occur between each dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04991532 — The tentative dosing schedule is 30, 100, 300, 600, 1200, and 2000 mg. Doses shown may be adjusted upwards or downwards and may be adjusted to include intermediate doses. All doses will be administered as extemporaneously-prepared powder in capsule (PIC) formulation.
  Arms: PF-04991532
Drug: Placebo — Placebo to match PF-04991532 will be provided
  Arms: Placebo

SUMMARY:
The purpose of this study is to characterize the safety, tolerability, pharmacokinetics (PK) and preliminary food effect of PF-04991532 following single escalating oral doses in healthy adult subjects.

DETAILED DESCRIPTION:
Safety/Tolerability and PK

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female (non child-bearing potential) subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 35.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
* Use of tobacco or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.
* Self-reported history of hypoglycemia, or fasting laboratory glucose value </=80 mg/dL at screening or Day 0 of Period 1, confirmed by a single repeat if deemed necessary.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability Endpoints: physical exams, AE monitoring, 12-lead ECGs, continuous cardiac monitoring, vital sign and clinical safety laboratory (including frequent glucose assessments via glucometer) measurements. | 1 month
PK Endpoints: AUC(0-inf), AUC(0-last), AUC(0-24), Cmax, Tmax, CL/F, Vz/F and half-life (t1/2), as the data permit. | 1 month

SECONDARY OUTCOMES:
none-see my comment

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2611001&StudyName=Single%20Dose%20Study%20of%20PF-04991532%20in%20Healthy%20Subjects